CLINICAL TRIAL: NCT02396472
Title: Internet Support Groups: Identifying and Improving Pathways for Mental Health
Brief Title: Mental Health Pathways in Internet Support Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Pittsburgh (Other); National Institute of Mental Health (NIMH) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: CarnegieMU
Record Dates: First submitted 2015-01-15; First posted 2015-03-24 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2019-08

CONDITIONS: Depression; Stress; Anxiety
Keywords: social support
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Order by time and topic (Placebo Comparator): Volunteers from the American Cancer Society's Cancer Survivors' Network (CSN) will see some of their messages delivered using CSN's default ordering, which shows messages within a conversational thread ordered by time stamp. Conversational threads are nested within a broad topic-based forum, like breast cancer or colorectal cancer survivors.
  Note that this is a within-participant trial, so that all participants participate in all arms of the trial. Messages, not people, are randomly assigned to condition.
  Interventions: Behavioral: Order by time and topic
- Order by information relevance (Active Comparator): In this condition some messages will be highlighted if they match the type of content the user has previously shown interest in, by previously contributing or reading semantically similar material.
  Interventions: Behavioral: Order by information relevance
- Order by social relationship (Active Comparator): In this condition some messages will be highlighted because they come from people the user has previously shown interest in, by previously reading their posts or communicating with them.
  Interventions: Behavioral: Order by social relationship
- Order by help giving (Active Comparator): In this condition some messages will be highlighted because they seek help and therefore provide an opportunity for participants to provide social support to others.
  Interventions: Behavioral: Order by help giving
- Order by self-disclosure (Active Comparator): In this condition some messages will be highlighted because in them the writer is self-disclosing, and they provide provide an opportunity for participants to self-disclose in return.
  Interventions: Behavioral: Order by self-disclosure

INTERVENTIONS:
Behavioral: Order by time and topic
  Arms: Order by time and topic
Behavioral: Order by information relevance
  Arms: Order by information relevance
Behavioral: Order by social relationship
  Arms: Order by social relationship
Behavioral: Order by help giving
  Arms: Order by help giving
Behavioral: Order by self-disclosure
  Arms: Order by self-disclosure

SUMMARY:
People facing serious health threats increasingly use Internet health support communities to obtain informational support, emotional support and other resources. This study introduces software algorithms similar to those used by social media sites to put people in touch with helpful information and social interactions. Participants from the American Cancer Society's Cancer Support Network will have access to this online support group using the default interface that orders content by broad content category and date or with a new interface that highlights communication content and people that match users' interests and needs.

DETAILED DESCRIPTION:
Internet support groups (ISGs) are online communities where people come together to exchange information, emotional support and other resources. They are an important resource for patients grappling with serious medical conditions. Although participation in health-related ISGs has been associated with significant reductions in participant-reported depression, anxiety and other indicators of psychological distress, many ISG members leave too soon to benefit. In a parallel study, we are using state-of-the art machine learning and automated language analysis techniques to assess the types of interactions that keep people participating in these groups and that lead to improved psychosocial well-being and health quality of life and how these interactions develop. The clinical trial described here uses these technologies and insights from our empirical research to build, deploy, and evaluate interventions that improve the interactions in Internet health support groups.

We will develop and pilot-test interventions to encourage effective communication processes identified in our empirical research. Participants from the American Cancer Society's Cancer Support Network will access this support group using either the default interface that orders content by disease diagnosis and date or with a new interface that sometimes highlights communication content and people who match their interests and needs. We will test whether mood, satisfaction with interactions and engagement in the group increase following interventions that (a) increase participants' receipt of individualized support from others; (b) provide participants with opportunities to offer support to others; (c) facilitate participants' expression of emotions; and (d) help participants form relationships with compatible peers. In a series of small, randomized experiments, we will examine how these interventions affect participants' communication behaviors as well as short-term engagement and satisfaction with their online interactions.

ELIGIBILITY:
Inclusion Criteria:

* Is an existing or new registrant to the American Cancer Society's Cancer Support Network.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6500 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Read message (Does the user read the message they were exposed to?) | 1 day

SECONDARY OUTCOMES:
Interaction satisfaction (Self-report measure of satisfaction 3-item survey) | 1 day
  Self-report measure of satisfaction with a random sample of messages. This is a 3-item survey that will be delivered as a pop-up questionnaire following a random sample of the messages users were exposed to.
Reply to message (How long does it take the users to reply to a message they were exposed to, if they reply at all.) | 2 days
  How long does it take the users to reply to a message they were exposed to, if they reply at all.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Kraut, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Wang YC, Kraut RE, Levine JM. Eliciting and receiving online support: using computer-aided content analysis to examine the dynamics of online social support. J Med Internet Res. 2015 Apr 20;17(4):e99. doi: 10.2196/jmir.3558. PMID 25896033
- [Background] Vlahovic, T., Wang, Y.-C., Kraut, R. E., & Levine, J. M. (2014). Support matching and satisfaction in an online breast cancer support community. CHI'14: Proceedings of the ACM Conference on Human Factors in Computing Systems (pp. 1625-1634 ). NY: ACM.
- [Background] Wang, Y., Kraut, R., & Levine, J. (2012). To stay or leave? the relationship of emotional and informational support to commitment in online health support groups CSCW '12 Proceedings of the ACM 2012 conference on Computer Supported Cooperative Work (pp. 833-842). NY: ACM.
- [Background] Yang D, Kraut R, Smith T, Mayfield E, Jurafsky D. Seekers, Providers, Welcomers, and Storytellers: Modeling Social Roles in Online Health Communities. Proc SIGCHI Conf Hum Factor Comput Syst. 2019 May;2019:344. doi: 10.1145/3290605.3300574. PMID 31423493
- [Background] Yang D, Yao Z, Seering J, Kraut R. The Channel Matters: Self-disclosure, Reciprocity and Social Support in Online Cancer Support Groups. Proc SIGCHI Conf Hum Factor Comput Syst. 2019 May;2019:31. doi: 10.1145/3290605.3300261. PMID 31448374
- [Background] Yang D, Yao Z, Kraut R. Self-disclosure and Channel Difference in Online Health Support Groups. Proc Int AAAI Conf Weblogs Soc Media. 2017 May;2017:704-707. PMID 31423352
- [Background] Yang D, Kraut R, Levine JM. Commitment of Newcomers and Old-timers to Online Health Support Communities. Proc SIGCHI Conf Hum Factor Comput Syst. 2017 May;2017:6363-6375. doi: 10.1145/3025453.3026008. PMID 31423492
- See also: Robert Kraut's recent articles and book chapters — https://kraut.hciresearch.info/articles/